CLINICAL TRIAL: NCT05812391
Title: Systemic Inflammatory Response Following Full Mouth Erythritol Powder Air Polishing and Instrumentation: A Randomized Clinical Trial
Brief Title: Impact of Full Mouth Erythritol Powder Air Polishing on Systemic Inflammatory Response
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Hayder Raad Abdulbaqi, Principal investigator, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Screening
Other Study IDs: 745622
Record Dates: First submitted 2023-04-02; First posted 2023-04-13 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Periodontal Diseases
Keywords: Periodontal disease; Periodontitis; Air abrasion; Tooth polishing; Air-polishing
MeSH Terms: conditions — Periodontal Diseases; Periodontitis | interventions — Congresses as Topic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test group (Active Comparator): Supra-gingival erythritol powerder air polishing Sub-gingival erythritol powerder air polishing Supra-gingival debridement Sub-gingival debridement
  Interventions: Procedure: test
- conventional group (Active Comparator): Supra-gingival debridement Sub-gingival debridement Polishing with polishing paste
  Interventions: Procedure: conventional

INTERVENTIONS:
Procedure: test — the treatment start with supra-gingival erythritol powerder air polishing followed by sub-gingival erythritol powerder air polishing,supra-gingival debridement and sub-gingival debridement
  Arms: test group
Procedure: conventional — the treatment start with supra-gingival debridement followed by sub-gingival debridement then finished with polishing paste
  Arms: conventional group

SUMMARY:
Periodontitis (PD) is an inflammatory condition that affects 20%-50% of the total global population, with severe disease occurring in 9.8% of individuals. clinically characterized by clinical attachment loss (CAL) and bleeding on probing (BOP) accompanied by increased probing pocket depth (PPD) and/or gingival recession, it may end with tooth loss if left untreated. non-surgical periodontal treatment (NSPT) represents the first line of treatment and involves the physical debridement of subgingival plaque biofilms. "full-mouth debridement" (FMD) approach, its NSPT delivers complete debridement within 24 hr. However, full-mouth NSPT has been consistently shown to trigger a large systemic inflammatory response 24 hr following treatment. Nevertheless, Interestingly, a positive correlation between treatment time and the subsequent systemic inflammatory response has been reported. Given this previous link and the different features of each instrumentation technique including air-polishing devices (APDs), that have less time-consuming treatment, reduce patient discomfort and sensitivity, and only minor alterations to surrounding soft and hard tissues. This study aims to evaluate the systemic inflammatory response following full-mouth erythritol powder air polishing and instrumentation.

DETAILED DESCRIPTION:
Periodontitis is a common chronic inflammatory disease caused by specific oral dysbiosis and characterized by a progressive loss of soft and hard tissues keeping the teeth. if left untreated, it leads not only to tooth loss, negative influences on the patient's quality of life and masticatory impairment may happen. There is significant evidence of clinical improvements in PD patients following non-surgical periodontal treatment (NSPT), including gains in clinical attachment level, reductions in gingival inflammation, and reduced periodontal pocket depths.

A conventional Full-mouth hand debridement has been consistently shown to trigger a large systemic inflammatory mediator, The reasons for such a response may be related to both the transient post-operative bacteremia and the extension of the operative trauma.

a recent joint consensus statement advised against full-mouth debridement for some medically compromised patients.

The erythritol powder is a water-soluble, non-toxic sugar alcohol and artificial sweetener, has a mean particle size of 14 μm, and can be used for supra and subgingival removal of biofilm and stains.

It has also been suggested that teeth with sites of furcation involvement and/or with reduced access, which have traditionally been difficult to debride with conventional instrumentation, may benefit from air-flow therapy

Comparing full-mouth ultrasonic debridement with polishing paste and full-mouth erythritol powder air polishing followed by ultrasonic debridement. this study hypothesized that the later procedure may reduce the extent of systemic inflammatory mediators they induce by removing the biofilm before the conventional full-mouth (supra and sub-gingival) ultrasonic debridement.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have periodontitis, unstable, at any stage

Exclusion Criteria:

* Participants who are known or suspected high risk for tuberculosis
* Participants who have hepatitis B or HIV infections
* Participants who are being unable to provide written, informed consent
* Participants who have history of bleeding diathesis
* Participants who are pregnant or intended to and lactating mother.
* Participants who are self-reported diagnosis of any systemic illnesses including cardiovascular, renal and liver diseases
* Participants who have regular use of medication to control systemic illness.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-03-10 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Change in serum level of C-reactive protein | 24 hours
  Change in serum level of C-reactive protein 24 hours following the full mouth debridement

SECONDARY OUTCOMES:
Treatment time | 30 days
  Evaluate the effect of treatment time (minute) on clinical parameters after 30 days
Change in percentage of bleeding on probing | 30 days
  Change in the percentage of bleeding on probing 30 days after treatment
Change in mean probing pocket depth | 30 days
  Change in mean probing pocket depth (mm) 30 days after treatment
Change in clinical attachment loss | 30 days
  Change in clinical attachment loss (mm)30 days after treatment
Change in percentage of plaque index | 30 days
  Change in percentage of plaque index 30 days after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed K Ayoob, Principal Investigator — University of Baghdad
Locations (1):
- Mohammed Kalid Ayoob, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No